CLINICAL TRIAL: NCT06133985
Title: Effects of Costovertebral Joint Mobilization on Respiratory Function in Asthmatic Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REC -01680 Bushra Ali Syed
Record Dates: First submitted 2023-10-25; First posted 2023-11-18 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2024-03

CONDITIONS: Asthmatic
Keywords: costovertebral joint mobilization; chest tightness; asthma; respiratory function
MeSH Terms: conditions — Asthma; Respiratory Aspiration

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Costovertebral mobilizations + Conventional Physiotherapy (Experimental): Costovertebral mobilizations along conventional treatment patient would receive costovertebral mobilization in side lying position for 10th to 6th ribs, in sitting position for 10th to 2nd rib and in supine position for 1 rib.
  Frequency: 5 times/week for 3 weeks. Intensity: moderate intensity (pain free) Time: 20 mins Type: costovertebral joint mobilization to improve respiratory function and chest tightness.
  Conventional treatment diaphragmatic breathing exercises and pursed-lip expiration exercises. Patient will receive diaphragmatic breathing and pursed lip breathing exercise in sitting position Frequency: 5 times/week for 3 weeks Intensity: moderate intensity (pain free) Time: 30 mins Type: breathing exercises to improve respiratory function and chest tightness.
  Interventions: Other: Costovertebral mobilizations + Conventional PT
- Conventional Physiotherapy (Other): diaphragmatic breathing exercises and pursed-lip expiration exercises Patient will receive diaphragmatic breathing and pursed lip breathing exercise in sitting position Frequency: 5 times/week for 3 weeks Intensity: moderate intensity (pain free) Time: 20 mins Type: breathing exercises to improve respiratory function and chest tightness.
  Interventions: Other: Conventional treatment

INTERVENTIONS:
Other: Costovertebral mobilizations + Conventional PT — Costovertebral mobilizations along conventional treatment patient would receive costovertebral mobilization in side lying position for 10th to 6th ribs, in sitting position for 10th to 2nd rib and in supine position for 1 rib.
  Frequency: 5 times/week for 3 weeks. Intensity: moderate intensity (pain free) Time: 10 mins Type: costovertebral joint mobilization to improve respiratory function and chest tightness.
  Conventional treatment diaphragmatic breathing exercises pursed-lip expiration exercises. Patient will receive diaphragmatic breathing and pursed lip breathing exercise in sitting position Frequency: 5 times/week for 3 weeks Intensity: moderate intensity (pain free) Time: 20 mins Type: breathing exercises to improve respiratory function and chest tightness.
  Arms: Costovertebral mobilizations + Conventional Physiotherapy
Other: Conventional treatment — diaphragmatic breathing exercises pursed-lip expiration exercises. Patient will receive diaphragmatic breathing and pursed lip breathing exercise in sitting position Frequency: 5 times/week for 3 weeks Intensity: moderate intensity (pain free) Time: 20 mins Type: breathing exercises to improve respiratory function and chest tightness.
  Arms: Conventional Physiotherapy

SUMMARY:
The aim of this randomized controlled trial is to determine the effectiveness of costovertebral joint mobilization on lung function in asthmatics. By targeting the thoracic region, costovertebral mobilization can play a valuable role in enhancing respiratory function and improving the overall well-being of individuals with respiratory conditions.

DETAILED DESCRIPTION:
Costovertebral joint mobilization can help to improve this by increasing the mobility of the ribs and thoracic spine, which can help to expand the chest and improve lung function. Additionally, costovertebral joint mobilization can help to reduce muscle tension in the chest and upper back, which can also contribute to improved respiratory function. This is because tense or tight muscles can restrict the movement of the rib cage, limiting the ability of the lungs to expand and contract. Mobilization are performed in three positions, sitting, supine lying and side lying with arm abducted of the side to be mobilized. The improvement by regular physical training of breathing technique and chest wall mechanics may be explained by mobilization of the costovertebral articulations.

ELIGIBILITY:
Inclusion Criteria:

* Force Expiratory Volume 1/Force Vital Capacity ratio less than 0.7
* Mild asthma (Force Expiratory Volume 1 over 70% predicted)
* Chest tightness (inspiratory muscle tightness)
* Altered Dyspnea index.

Exclusion Criteria:

* presence of any underlying lung condition other than asthma.
* significant cardiovascular or musculoskeletal disease that may compromise the participant's capacity to participate in physical activity;
* active cancer.
* uncontrolled hypertension or diabetes.

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2023-10-01 (Actual); Primary Completion 2024-02-01 (Actual); Study Completion 2024-02-01 (Actual)

PRIMARY OUTCOMES:
Assessment of respiratory function FEV1 using spirometer. | 3 weeks
  Spirometry is one of the Pulmonary Function Test; they are useful investigations in the management of patients with respiratory disease or respiratory weakness secondary to neurological impairment. Spirometry will measure FEV1
Assessment of respiratory function FVC using spirometer. | 3 weeks
  Spirometry is one of the Pulmonary Function Test; they are useful investigations in the management of patients with respiratory disease or respiratory weakness secondary to neurological impairment. Spirometry will measure FVC
Tape for chest expansion | 3 weeks
  Chest expansion is measured using a measuring tape at 2 different levels of the rib cage. The 2 measurements of chest diameter are taken at the end of deep inspiratory and expiratory maneuvers. Upper and lower chest expansion are obtained by subtracting the inspiratory diameter from the expiratory diameter, according to the designated anatomical markers. The assessment is performed 1 measurement of upper chest expansion and then 1 measurement of the lower chest expansion consecutively, holding the measuring tape at both ends with thumb and index finger around the patient body.
Dyspnea index | 3 weeks
  It is used to describe their sense of breathlessness and breathing problem, and the effects of their breathing on their lives.

CONTACTS AND LOCATIONS:
Overall Officials: Asghar Khan, DPT,DSc PT, Principal Investigator — Riphah International University
Locations (1):
- Rahim Hospital, Rawalpindi, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No